CLINICAL TRIAL: NCT05763888
Title: An Exploratory Approach for Validation and Standardization of Test Methods and Evaluators to Conduct In-Vivo Clinical Safety and Efficacy Testing of Hair Care Range of Products
Brief Title: Validation and Standardization of Test Methods and Evaluators for Testing of Hair Care Range of Products
Status: Completed | Type: Observational
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Principal Investigator, Maheshvari Patel, Principal Investigator, NovoBliss Research Pvt Ltd
Other Study IDs: NB220039-NB
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Healthy Subject

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No drug will given — No intervention will be given to the subject

SUMMARY:
An exploratory approach for validation and standardization of test methods and evaluators to conduct In-Vivo clinical safety and efficacy testing of hair care range of products.

A total of 40 subjects will be enrolled.

DETAILED DESCRIPTION:
This is an internal standardization and validation study. This standardization and validation study will be carried out by the trainee evaluators' of NovoBliss Research who voluntarily wish to take part in this study. There are multiple techniques for establishing documentary evidence demonstrating that standardised procedural steps, processes and methods are carried out in testing for hairs care range of products to maintain the desired level of compliance.

It is very important that in addition to final testing and compliance of products, it is also assured that the process will consistently produce the expected results. The desired results are established in terms of specifications for the outcome of the processes.

Below listed test methods/techniques will be performed:

* Assessment of General appearance of hair (i.e. Hair Volume, Hair Density, Hair Reflection, Hair Plasticity, Hair Smoothness, Hair Oiliness, Shininess)
* Assessment of Scalp Appearance i.e. itchiness, dryness, redness, roughness, and scaliness of scalp
* Assessment of Adherent Scalp Flaking Score (ASFS)
* Assessment of Hair Strength (i.e. Poor, Average, Good)
* Assessment of Gray Hair - Graying Severity Score (GSS); Hair Whitening Score. Evaluation Methods
* 60-seconds hair count (Hair Combing Method)
* Hair Pull Test
* Trichogram (Pluck Test - Anagen: Telogen Ratio Calculation)
* Scanning Electron Microscope (SEM)

Instrumental Evaluation:

* Phototrichogram - Tattoo Method for Hair Growth Rate, Hair Density, Hair Thickness, and Scalp Condition i.e. Scalp Dandruff - Using CASLite Nova
* Scalp Hydration by MoistureMeterEpiD
* Scalp Sebum level by Sebumeter
* Hair Color by Hair/Skin Colorimeter CL 410
* Image analysis for Hair Growth Rates, number of hairs and length, and Gray hair counts, using Image-Pro Software
* Assessment of Hair Cuticle - by Electron microscope to check parameters such as surface damage of hair, photodamage of outermost cuticle layer
* Microbial changes in scalp flora by trichoscopy or dermoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 75 years (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Females of childbearing potential must have a self-reported negative urine pregnancy.
4. Subject is in good general health as determined by the Investigator on the basis of medical history.
5. Subject is willing and able to follow and allow study staff to performed study test methods
6. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
7. Subject must be able to understand and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Subject have history of allergy to any ink.
2. Subject have participated any clinical research study related to hair care products.
3. Subject having history of diabetes
4. Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.
5. Subject having known history of any skin diseases including eczema, atopic dermatitis or active cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Referring to the convenience sampling method which is a type of non-probability sampling, a total of 40 subjects will be enrolled. This technique involves selecting a research sample based on convenience & accessibility, drawing the sample from the part of the population close to hand.
  In this study, the purpose is to standardize and validate the methods and evaluators' and there is no usage of medicines/test articles/test treatment or test products, specific sample calculation of sample size estimation is not required.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the standardize the methods, procedural steps | Day 01 to Day 04
  Validate the hair growth rate measurement
Evaluate the standardize the methods, procedural steps | Day 01 to Day 04
  60-s combing test
Evaluate the standardize the methods, procedural steps | Day 01 to Day 04
  Hair Pull test
Evaluate the standardize the methods, procedural steps | Day 01 to Day 04
  Hair Pluck test
Evaluate the standardize the methods, procedural steps | Day 01 to Day 04
  Subjective scoring of Hair quality appearance and scalp condition

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, MBBS, Study Director — Medical Director
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No